CLINICAL TRIAL: NCT06949319
Title: Individualized Stroke Risk Scores and Hemostatic Profile in Oral Anticoagulant-naïve (OAC-naïve) Patients With Non-valvular Atrial Fibrillation (NVAF)
Brief Title: Stroke Risk Assessment and Markers of Blood Clotting in Patients With Newly Diagnosed Non-valvular Atrial Fibrillation (NVAF), Who Have Not Received Oral Anticoagulation Therapy (OAC-therapy) Prior to Inclusion
Acronym: BIO-AF
Status: Recruiting | Type: Observational
Sponsor: Nedim Tojaga (Other)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other); Karola Jørgensens Foundation and Foundation for Cardiology in Southwest Denmark. (Unknown); Grosserer L.F. Foghts Foundation (Unknown); Direktør Kurt Bønnelycke og Hustru fru Grethe Bønnelyckes Fond (Unknown); The Faculty of Health Sciences SDU (Unknown); Research Electronic Data Capture (REDCap) (Unknown); Region of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Nedim Tojaga, Principal investigator., University of Southern Denmark
Organization: University of Southern Denmark (Other)
Other Study IDs: S-20240018
Record Dates: First submitted 2025-02-05; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation (Prevention of Stroke); Atrial Fibrillation New Onset; Non Valvular Atrial Fibrillation; Stroke (in Patients With Atrial Fibrillation); Stroke; Thrombosis
Keywords: Stroke risk assessment in patients with atrial fibrillation; OAC-naïve patients with newly diagnosed atrial fibrillation; Hemostatic biomarkers; CHA2DS2-VASc score; ABC-stroke score; AF-burden; Left Atrial Function Index (LAFI); Echocardiography; HFA-PEFF score; H2FPEF score; Heart failure with preserved ejection fraction (HFpEF); Stroke; Oral anticoagulant therapy; Non-valvular atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fasting blood samples will be drawn from an antecubital vein with minimal stasis, using a 21 gauge needle. The first 2 mL of blood will be discarded, and the following 6 x 2.7 mL blood will be collected into 0.109 M sodium citrate tubes for APTT, INR, and hemostasis variables. Then, 2 x 3 mL of blood will be collected in Li-Heparin tubes for lipids, liver enzymes, renal function, CRP, NT-proBNP, and hs-TNT. Finally, 3 mL of blood will be collected in EDTA-tubes for HbA1c and full blood count. To generate platelet poor plasma (PPP), the tubes will be centrifuged at 2000 g for 20 min. at room temperature. PPP will be stored at -80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oral anticoagulant-naïve (OAC-naïve) patients with non-valvular atrial fibrillation (NVAF).: The study population will consist of patients with newly diagnosed non-valvular atrial fibrillation (NVAF). Patients will have to be naïve to oral and parenteral anticoagulants prior to inclusion. Patients with newly diagnosed NVAF who are willing to participate in this study and sign the patient consent form will be scheduled for fast track outpatient clinic visit within four days for blood sampling, transthoracic echocardiography (TTE), and heart rhythm monitoring. OAC treatment will be initiated immediately after blood sampling, based on current guidelines for the management of NVAF. Demographic data will be collected, as well. Likewise, symptoms attributable to NVAF will be quantified according to the modified EHRA-score (European Heart Rhythm Association). Investigators will also determine whether hypertension and diabetes are effectively managed by home blood pressure (BP) measurements and HbA1c levels.

SUMMARY:
Background:

Atrial fibrillation (AF) is the most common heart rhythm disorder worldwide. Globally, there are 37.5 million people with AF. AF increases the risk of death, heart failure, and stroke, which severely affect patients and also lead to high healthcare costs. Around 25% of all strokes are caused by AF, and patients with stroke due to AF tend to have a higher risk of death and more disability compared to stroke patients without AF.

Stroke prevention is, therefore, an important part of AF treatment, in which blood thinning medication has an important role. However, blood thinners increase the risk of bleeding. Therefore, it is important to divide patients with AF into different risk groups, known as risk assessment, to figure out who will benefit the most from blood thinners. To be able to divide patients into different risk groups, various stroke risk assessment tools have been developed, such as the CHA2DS2-VASc score and the ABC-stroke score. The most commonly used tool is the CHA2DS2-VASc score, including only clinical risk factors, such as high blood pressure, diabetes, etc. The ABC-stroke score, which includes blood markers of heart function, has been proven to outperform the CHA2DS2-VASc score in terms of predicting stroke in AF patients. However, the CHA2DS2-VASc score remains the primary stroke risk assessment tool for AF patients in current guidelines.

After looking at the different risk factors, patients are divided into three groups: low, intermediate, and high risk. High-risk patients must take blood-thinning medication for life, while low-risk patients do not need it. In the medium-risk group, it remains uncertain whether blood thinners should be given or not.

Despite the broad use of the CHA2DS2-VASc score, the score itself has limitations. The score does not include important factors, such as the duration of AF, the size and function of the upper heart chambers, as well as the stiffness of the heart, and markers of blood clotting, which are proven markers of a state that inceases the risk of blood clots. Furthermore, the CHA2DS2-VASc score does not consider whether heart failure, high blood pressure, and diabetes are well-controlled or not, which could lead to overuse of blood thinners. Therefore, the current risk assessment tools for patients with AF are incomplete, and improvements are needed.

Overall hypothesis:

Overall hypothesis is that the different components of the CHA2DS2-VASc score and ABC-stroke score affect blood clotting markers differently, depending on whether conditions like heart failure, high blood pressure, and diabetes (modifiable risk factors) are well-controlled or not. Investigators also expect to see differences in blood clotting markers across different stroke risk groups (low, intermediate, and high risk, based on the CHA2DS2-VASc score and ABC-stroke score) in AF patients who have not yet started blood thinning medication. Furthermore, investigators believe that the duration of AF, the size/function of the upper heart chambers, as well as the stiffness of the heart, can reflect an increased risk of blood clots in AF patients.

Overall goal of the study:

The overall goal of the study is to help improve the current tools used to assess the risk of stroke in patients with newly diagnosed AF. This will be done by adding more factors to the current risk assessment tools that reflect an increased risk of stroke, such as the burden of AF, the size/function of the heart's upper chambers, as well as the stiffness of the heart, and using biomarkers that show the blood's ability to clot as a substitute measure for stroke risk.

Methods:

The study is a cross-sectional, single-center observational study and will take place at Esbjerg Hospital - University Hospital of Southern Denmark, involving collaboration between the Unit for Thrombosis Research, Department of Clinical Diagnostics and the Department of Cardiology.

The study population will consist of 150 participants with newly diagnosed AF. The participants must not be taking a specific type of blood thinner, called anticoagulant therapy (OAC-therapy), before being included in the study. The participants will be recruited with the help of the general practitioners (GPs). The general practitioners will be thoroughly informed about the study and the importance of waiting to start OAC-therapy until the participants have been seen at the cardiology outpatient clinic. The participants will be scheduled for a blood test, an ultrasound of the heart (echocardiography), and a 7-day heart rhythm monitoring within 4 days after their first meeting with the GP.

DETAILED DESCRIPTION:
Background:

Non-valvular atrial fibrillation (NVAF) is the most prevalent cardiac arrhythmia worldwide, and it is associated with a five-fold increased risk of ischemic stroke compared to a healthy population. Patients with stroke due to atrial fibrillation (AF) have a higher mortality and greater disability compared to stroke patients without AF.

Oral anticoagulants (OACs), either vitamin K antagonists (VKAs) or direct oral anticoagulants (DOACs), are the cornerstones for the prevention of ischemic strokes in patients with AF. Different stroke risk stratification schemes have been developed to guide OAC therapy decision-making in AF patients. The most commonly used scheme is the CHA2DS2-VASc score, including the clinical risk factors congestive heart failure, hypertension, age, diabetes, prior stroke, vascular disease, and female gender. One point is assigned for every risk factor encompassed by the CHA2DS2-VASc score, except age ≥75 years and prior stroke, which account for two points each. The score ranges from 0-9 points, with higher scores representing a higher risk of stroke. The annual risk of ischemic stroke for CHA2DS2-VASc score of 0, 1, and 2 is approximately 0-0.68 %, 1.3-1.61 %, and 2.2-2.49 %, respectively. Novel stroke risk stratification schemes, also incorporating biomarkers, have been developed, e.g., the ABC-stroke score (Age, Biomarkers, and Clinical history). The components of the ABC-stroke score include age, plasma levels of N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) and high-sensitivity troponin T (hs-TNT), and prior stroke/transient ischemic attack (TIA). ABC-stroke risk categories are defined as low-risk (<1 % predicted one-year risk of stroke), medium-risk (1-2 % predicted one-year risk of stroke), and high-risk (>2 % predicted one-year risk of stroke). Studies have shown that the ABC-stroke score outperforms the CHA2DS2-VASc score in terms of stroke risk prediction and stratification of AF patients. However, the CHA2DS2-VASc score is still recommended as the primary stroke risk stratification scheme for AF patients in current guidelines. Despite the broad use of stroke risk stratification schemes in clinical practice, stroke risk assessment remains particularly challenging in AF patients with intermediate stroke risk, i.e., men with a CHA2DS2-VASc score of 1 and women with a CHA2DS2-VASc score of 2, where current guidelines recommend considering OAC therapy. OAC therapy is generally recommended for AF patients at high risk of stroke, i.e., men with CHA2DS2-VASc score of ≥ 2 and women with CHA2DS2-VASc score of ≥ 3. OAC therapy is generally not recommended for AF patients at low risk of stroke, i.e., men with a CHA2DS2-VASc score of 0 and women with a CHA2DS2-VASc score of 1.

The CHA2DS2-VASc score is broadly used in clinical practice due to its simplicity and low cost, however, the score has limitations. It exclusively includes clinical stroke-related risk factors, but not AF burden and left atrial size/function, which are proven independent markers of a hypercoagulable state. Treatment and stroke risk assessment in AF patients is moving towards a more individualized patient care, in which biomarkers play an essential role in improving risk stratification and personalizing treatment, as proposed in the ABC-stroke score. In recent years, measurements of hemostatic biomarkers in AF patients have been investigated in several studies, illustrating a hypercoagulable state. Of note, the CHA2DS2-VASc score also predicts stroke risk in patients without AF. Hence, there are concerns about the specificity for predicting AF-related stroke versus non-AF related stroke. Furthermore, the CHA2DS2-VASc score does not consider whether the modifiable components are well-controlled or not, which could lead to OAC overtreatment. For these reasons, there is still a need for refining stroke risk prediction using more AF-sensitive factors (i.e., AF-burden and left atrial size/function), in addition to the clinical factors, and for more exhaustive assessment of the modifiable components, to optimize stroke risk stratification in the future. It remains to be established whether the abovementioned AF-sensitive factors can be used to improve OAC decision-making, particularly in NVAF patients with intermediate stroke risk, where the balance between benefit and harm is less clear. When doubt persists, the presence of one or more non-CHA2DS2-VASc stroke risk factors could possibly strengthen the decision to initiate OAC therapy.

The annual risk of ischemic stroke in NVAF patients depends on the overall CHA2DS2-VASc score. However, the annual risk of ischemic stroke in patients with NVAF may differ depending on the individual components of the CHA2DS2-VASc score that determine the score, despite the overall score being the same, as well as whether the modifiable components are well-controlled or not. Glowicki et al. conducted a study comparing the hemostatic profiles of AF patients with low stroke risk to those with intermediate stroke risk, as determined by the CHA2DS2-VASc score. As opposed to the study by Glowicki et al., this study will compare all three stroke risk groups, i.e., low, intermediate, and high risk, as determined by the CHA2DS2-VASc score and ABC-stroke score, and will incorporate a broader panel of hemostatic biomarkers, including the contact activation system. Furthermore, this study will investigate AF-burden and left atrial size/function, and their association with the hemostatic profile. Patients included in this study will be genuinely OAC-naïve, as opposed to the study by Glowicki et al. Comparison of hemostatic profiles between different stroke risk groups could be essential for the future improvement of OAC therapy decision-making, especially in NVAF patients with intermediate stroke risk.

Objectives:

* To evaluate how the individual components of the CHA2DS2-VASc score and ABC-stroke score are associated with hemostatic biomarkers, including an assessment of whether the modifiable components are well-controlled or not, and how the hemostatic profile differs among stroke risk groups in OAC-naïve NVAF patients.
* To compare the hemostatic profiles of the different CHA2DS2-VASc scores and ABC-stroke scores in OAC-naïve NVAF patients.
* To evaluate how AF-burden is associated with hemostatic biomarkers in OAC-naïve NVAF patients.
* To evaluate how left atrial size/function is associated with hemostatic biomarkers in OAC-naïve NVAF patients.
* To evaluate how underlying heart failure with preserved ejection fraction (HFpEF) is associated with hemostatic biomarkers in OAC-naïve NVAF patients.

Materials and methods:

Study Design: The study consists of five substudies. The first substudy will investigate the association of the different CHA2DS2-VASc score and ABC-stroke score components with the hemostatic profile in OAC-naïve NVAF patients. Furthermore, assessment of whether the modifiable components of the CHA2DS2-VASc score (i.e., diabetes and hypertension) are well-controlled or not, and its impact on the hemostatic profile will be investigated. Likewise, the hemostatic profile of OAC-naïve NVAF patients with intermediate stroke risk will be compared to that of OAC-naïve NVAF patients with low and high stroke risks, respectively, to determine which of the two groups most closely resembles patients with intermediate stroke risk in terms of their hemostatic profile. The second substudy will compare the hemostatic profile between the CHA2DS2-VASc score and ABC-stroke score in OAC-naïve NVAF patients. The third substudy will investigate how AF-burden is associated with hemostatic biomarkers in OAC-naïve NVAF patients. AF-burden will be determined as a percentage based on the total number of AF-events during seven days heart rhythm monitoring. In the fourth substudy, investigators will evaluate how left atrial size/function is associated with hemostatic biomarkers in OAC-naïve NVAF patients. In the fifth substudy, investigators will investigate how underlying HFpEF is associated with hemostatic biomarkers in OAC-naïve NVAF patients. HFpEF will be evaluated using the HFA-PEFF and H2FPEF scores. The study is a cross-sectional, single-center observational study and will take place at Esbjerg Hospital - University Hospital of Southern Denmark, involving collaboration between the Unit for Thrombosis Research, Department of Clinical Diagnostics and the Department of Cardiology.

Study population: The study population will consist of patients with newly diagnosed NVAF. Patients will have to be naïve to oral and parenteral anticoagulants prior to inclusion. Investigators will check for this upon inclusion by systematic screening of an online medication database, called FMK, which is widely used among health care personnel in Denmark. According to the annual report (2023) from the AF database in Denmark (AFDK), there are about 800 patients with newly diagnosed AF in the catchment area of the University Hospital of Southern Denmark, Esbjerg, why investigators are confident that it will be possible to include the necessary number of patients. Collaboration with the general practitioners will be essential for patient inclusion. Investigators will provide comprehensive information to general practitioners about this study and the importance of withholding OAC treatment before subacute referral to the Department of Cardiology. Patients with newly diagnosed NVAF who are willing to participate in this study and sign the patient consent form will be scheduled for fast track outpatient clinic visit within four days of their consultation with the general practitioner for blood sampling, transthoracic echocardiography (TTE), and heart rhythm monitoring. OAC treatment will be initiated immediately after blood sampling, based on current guidelines for the management of AF, and investigators will also do a tailored comprehensive work-up of the AF patients as necessary. Demographic data will be collected, as well. Likewise, symptoms attributable to AF will be quantified according to the modified EHRA-score (European Heart Rhythm Association). To exclude other causes of coagulopathy and characterize the patients at baseline, investigators will measure the following variables in each participant: Full blood count, Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR), renal function, Glycated Hemoglobin (HbA1c), C-reactive Protein (CRP), liver function, and lipid profiles. Furthermore, plasma levels of NT-proBNP and hs-TNT will be determined with high-sensitivity immunoassays to estimate the ABC-stroke score. The risk of thromboembolic events will be estimated using the CHA2DS2-VASc score and ABC-stroke score for all patients in this study population, and the patients will be grouped according to their overall individual score. Moreover, each group will be subdivided according to the individual components of the CHA2DS2-VASc score and ABC-stroke score that constitute the overall score. Investigators will determine whether hypertension and diabetes are effectively managed by conducting home blood pressure (BP) measurements and assessing HbA1c levels. BP will be measured at home three times in the morning and evening over three consecutive days, and mean BP will be calculated based on the measurements from days two and three. For simplicity, well-controlled hypertension will be defined as a BP ≤ 135/85 mmHg, and a systolic BP ≤ 145 mmHg for age groups < 80 years and ≥ 80 years, respectively. The treatment goals for type 1 and 2 diabetes patients are HbA1c ≤ 53 and ≤ 48 mmol/mol, respectively, and will be used as thresholds for whether diabetes is well controlled or not.

Sample size estimation and statistical analyses: For sample size calculation, investigators utilized the median values and interquartile ranges of endogenous thrombin potential (ETP), as previously compared between AF patients with low and intermediate stroke risk by Glowicki et al. If the true difference of ETP between the low and intermediate stroke risk means is 120 nmol/L x min., and if investigators want to achieve power of 80 %, the sample size of the smallest group needs to contain at least 18 patients. According to the annual report (2023) from AFDK, approximately 12 % of incident AF patients in the Region of Southern Denmark were low-risk, 30 % were intermediate-risk, and 58 % were high-risk, as estimated by the CHA2DS2-VASc score. Given this distribution, investigators would need 150 AF patients in the overall study population to be able to answer whether ETP differs between the three stroke risk groups, i.e., low-risk, intermediate-risk, and high-risk groups. Investigators will use analysis of variance (Anova) to compare the three different stroke risk groups. Pearson's correlation or Spearman's rank correlation will be used to assess correlations between components of the CHA2DS2-VASc and ABC-stroke scores, AF-burden, left atrial size/function, and hemostatic biomarkers. A P-value <0.05 will be considered statistically significant.

Blood sampling: Fasting blood samples will be drawn from an antecubital vein with minimal stasis, using a 21 gauge needle. The first 2 mL of blood will be discarded, and the following 6 x 2.7 mL blood will be collected into 0.109 M sodium citrate tubes for APTT, INR, and hemostasis variables. Then, 2 x 3 mL of blood will be collected in Li-Heparin tubes for lipids, liver enzymes, renal function, CRP, NT-proBNP, and hs-TNT. Finally, 3 mL of blood will be collected in EDTA-tubes for HbA1c and full blood count. To generate platelet poor plasma (PPP), the tubes will be centrifuged at 2000 g for 20 min. at room temperature. PPP will be stored at -80°C until analysis.

Hemostatic biomarkers: Investigators will measure biomarkers related to the primary and secondary hemostasis, as listed below:

Primary hemostasis (platelet plug formation): To assess the influence of the primary hemostasis, investigators will measure the levels of von Willebrand factor (vWF) antigen using an in-house enzyme-linked immunosorbent assay (ELISA). If the concentrations of vWF are elevated compared with reference values, p-selectin and ADAMTS13 will be analyzed.

Secondary hemostasis (fibrin formation and resolution): Assessment of the secondary hemostasis will be done by analyzing thrombin turnover, and investigate whether thrombin generation is initiated though the contact activation system (CAS), i.e., the intrinsic pathway of the coagulation cascade, or the tissue factor (TF) pathway, i.e., the extrinsic pathway. In relation to CAS, measures of kallikrein generation (lag time, peak kallikrein concentration, time to peak, and endogenous kallikrein potential (EKP)) and concentrations of cleaved high-molecular weight kininogen (cHK), factor XII, prekallikrein, and HK will be measured. Concentrations of C1-inhibitor will be measured with commercial C1-inhibitor antibodies. Thrombin generation will be assessed through measures of lag time, peak thrombin concentration, time to peak, and endogenous thrombin potential (ETP). Endogenous activation of prothrombin to thrombin will be estimated from concentrations of prothrombin fragment 1 + 2 (F1+2), by a commercial ELISA. Furthermore, factor VII, factor X, factor II, protein C, protein S, tissue factor pathway inhibitor (TFPI), and antithrombin (AT) will be measured using commercial ELISAs to assess concentrations of activators and inhibitors of blood coagulation. Fibrin turnover will be assessed through fibrin clot lysis and concentrations of fibrinogen, which will be measured on a BN II analyzer. To assess fibrinolysis, D-dimer, a fibrin degradation product, will be measured by an immunoturbidimetric method. Other markers of fibrinolysis will be measured as well, i.e., tissue-type plasminogen activator (t-PA), plasminogen activator inhibitor 1 (PAI-1), plasminogen, plasmin inhibitor (PI), factor XIII, and thrombin activatable fibrinolysis inhibitor (TAFI), using in house and commercial assays.

AF burden, left atrial function, and HFpEF: Participants will undergo transthoracic echocardiography (TTE) as well as seven days heart rhythm monitoring. Through TTE, a rhythm independent expression of left atrial function, known as left atrial function index (LAFI), will be calculated. LAFI is a ratio that incorporates analogues of cardiac output, atrial reservoir function, and left atrial (LA) size. It is calculated as LAFI = (LA Emptying Fraction (LAEF) x Left Ventricular Outflow Tract - Velocity Time Integral (LVOT-VTI))/LA End-Systolic Volume Index (LAESVI). LAEF is the difference between LA end-systolic volume (LAESV) and LA end-diastolic volume (LAEDV) divided by LAESV and multiplied by 100, which is illustrated as LAEF = ((LAESV-LAEDV)/LAESV) x 100. LVOT-VTI is calculated by placing the pulsed wave doppler sample volume in the LVOT below the aortic valve and trace the velocity curves. LVOT-VTI is expressed in cm and describes the distance blood travels in one heartbeat. LAESVI is the largest LA volume in end-systole in mL indexed to body surface area (BSA). Left atrial function has been proven to modify the risk of stroke in patients with NVAF. Left Ventricular Ejection Fraction (LVEF) will also be assessed as part of the TTE. Furthermore, echocardiographic assessment of underlying HFpEF will be made through the HFA-PEFF score and the H2FPEF score. AF-burden will be determined as a percentage based on the total number of AF-events during the seven days heart rhythm monitoring. This is of prognostic importance due to growing evidence indicating a substantial association between AF burden and stroke.

Primary and secondary endpoints: Studies have shown that activation of the coagulation cascade (secondary hemostasis) is the most significant cause of a prothrombotic state, for which thrombin plays an essential role. Therefore, primary endpoints will be related to thrombin generation, kallikrein generation, and F1 + 2. Secondary endpoints will be the remaining hemostatic biomarkers, AF-burden, LAFI, and underlying HFpEF.

Ethical considerations:

Participants will be meticulously informed about this study, and all questions paticipants might have will be answered. Participants will have to sign the patient consent form prior to enrollment. Data will be stored in a secure database, in accordance with Danish and European legislation. In general, this research will be conducted in accordance with the Declaration of Helsinki.

Clinical relevance:

OAC therapy plays an essential role in stroke risk reduction in patients with AF. The CHA2DS2-VASc score is used in everyday clinical practice to determine the potential need for OAC therapy in patients with AF. However, novel stroke risk stratification schemes incorporating biomarkers have been developed, e.g., the ABC-stroke score, which has been shown to outperform the CHA2DS2-VASc score, in terms of stroke risk prediction and stratification of AF patients. It remains unknown how the individual components of the CHA2DS2-VASc score and ABC-stroke score affect the hemostatic profile in patients with NVAF, and how the hemostatic profile differs among stroke risk groups. Furthermore, the CHA2DS2-VASc score does not consider whether the modifiable components are well-controlled or not, which could possibly lead to OAC overtreatment. Likewise, the CHA2DS2-VASc score and ABC-stroke score do not account for key factors (e.g., AF-burden and left atrial size/function) that are able to impact stroke event rates. The lack of abovementioned factors is believed to be a major limitation of the CHA2DS2-VASc score, in particular. Investigators believe that using AF-burden and left atrial size/function in addition to the CHA2DS2-VASc score and ABC-stroke score could improve OAC decision-making, especially in NVAF patients with intermediate stroke risk. The first step is to characterize the CHA2DS2-VASc score/ABC-stroke score, AF-burden, and left atrial size/function with respect to the hemostatic profile. In this way, this study lays the foundation for future prospective studies investigating whether adding non-clinical factors to the CHA2DS2-VASc score and ABC-stroke score can improve stroke risk stratification in OAC-naïve NVAF patients.

Impact paragraph:

AF accounts for 25 % of ischemic strokes. Stroke can cause long-term disability and remains the second leading cause of death worldwide. OAC therapy is important for stroke prevention in AF patients. The CHA2DS2-VASc score and ABC-stroke score are used for stroke risk stratification and OAC therapy decision-making in AF patients. However, the CHA2DS2-VASc score, in particular, is associated with limitations, i.e., lack of AF sensitive factors. This study will, through the use of AF-burden and left atrial size/function, in addition to the CHA2DS2-VASc score and ABC-stroke score, seek to lay the foundation for future improvement of OAC therapy decision-making, particularly in NVAF patients with intermediate stroke risk. Investigators believe that this project is in line with UN's sustainable development goal number three (i.e., good health and well-being) due to contributing to stroke risk stratification advances in OAC-naïve NVAF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed non-valvular atrial fibrillation (NVAF), who are oral anticoagulant-naïve (OAC-naïve) prior to inclusion.
* Age ≥ 18 years.
* Signed informed consent.

Exclusion Criteria:

* Ongoing OAC treatment prior to inclusion.
* Valvular AF (mechanical heart valves or moderate-severe mitral stenosis).
* Secondary AF due to an acute reversible precipitant (e.g., infection, surgery, thyrotoxicosis, etc.).
* Pregnant or breastfeeding women.
* Treatment with oral contraceptives.
* End-stage renal disease (creatinine clearance <15 mL/min as calculated by the Cockcroft-Gault equation).
* Connective tissue diseases.
* Active cancer (cancer diagnosis not followed by curative procedures six months from the date of diagnosis).
* Major surgery (< three months).
* Acute coronary syndrome, stroke/TIA, and venous thromboembolism within three months prior to inclusion.
* Thrombophilia.
* Significant liver disease.
* Significant hematological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with newly diagnosed non valvular atrial fibrillation (NVAF). Patients will have to be naïve to oral and parenteral anticoagulants prior to inclusion. Study participants will be enrolled from the catchment area of the University Hospital of Southern Denmark, Esbjerg. Collaboration with the general practitioners will be essential for patient inclusion. Investigators will provide comprehensive information to general practitioners about this study and the importance of withholding OAC treatment before subacute referral to the Department of Cardiology. Patients with newly diagnosed NVAF who are willing to participate in this study and sign the patient consent form will be scheduled for fast track outpatient clinic visit within four days of their consultation with the general practitioner for blood sampling, transthoracic echocardiography (TTE), and heart rhythm monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Thrombin generation assessed by lag time | Thrombin generation, assessed by lag time, will be measured at baseline (enrollment).
  Thrombin generation plays a pivotal role in blood clotting and thus serve as primary outcome measure. Thrombin generation will be assessed through measurement of lag time (min), using the calibrated automated thrombography (CAT) method.
Thrombin generation assessed by peak thrombin concentration | Thrombin generation, assessed by peak thrombin concentration, will be measured at baseline (enrollment).
  Thrombin generation plays a pivotal role in blood clotting and thus serve as primary outcome measure. Thrombin generation will be assessed through measurement of peak thrombin concentration (nmol/L), using the calibrated automated thrombography (CAT) method.
Thrombin generation assessed by time to peak | Thrombin generation, assessed by time to peak, will be measured at baseline (enrollment).
  Thrombin generation plays a pivotal role in blood clotting and thus serve as primary outcome measure. Thrombin generation will be assessed through measurement of time to peak (min), using the calibrated automated thrombography (CAT) method.
Thrombin generation assessed by endogenous thrombin potential | Thrombin generation, assessed by endogenous thrombin potential, will be measured at baseline (enrollment).
  Thrombin generation plays a pivotal role in blood clotting and thus serve as primary outcome measure. Thrombin generation will be assessed through measurement of endogenous thrombin potential (nmol/L x min), using the calibrated automated thrombography (CAT) method.
Kallikrein generation assessed by lag time | Kallikrein generation, assessed by lag time, will be measured at baseline (enrollment).
  Kallikrein generation plays an important role in the contact activation system of the secondary hemostasis, therefore it will serve as a primary outcome measure. Kallikrein generation will be assessed through measurement of lag time (min), using the calibrated automated thrombography (CAT) method.
Kallikrein generation assessed by peak kallikrein concentration | Kallikrein generation, assessed by peak kallikrein concentration, will be measured at baseline (enrollment).
  Kallikrein generation plays an important role in the contact activation system of the secondary hemostasis, therefore it will serve as a primary outcome measure. Kallikrein generation will be assessed through measurement of peak kallikrein concentration (nmol/L), using the calibrated automated thrombography (CAT) method.
Kallikrein generation assessed by time to peak | Kallikrein generation, assessed by time to peak, will be measured at baseline (enrollment).
  Kallikrein generation plays an important role in the contact activation system of the secondary hemostasis, therefore it will serve as a primary outcome measure. Kallikrein generation will be assessed through measurement of time to peak (min), using the calibrated automated thrombography (CAT) method.
Kallikrein generation assessed by endogenous kallikrein potential | Kallikrein generation, assessed by endogenous kallikrein potential, will be measured at baseline (enrollment).
  Kallikrein generation plays an important role in the contact activation system of the secondary hemostasis, therefore it will serve as a primary outcome measure. Kallikrein generation will be assessed through measurement of endogenous kallikrein potential (nmol/L*min), using the calibrated automated thrombography (CAT) method.
Concentrations of prothrombin fragment 1 + 2 | Prothrombin fragment 1 + 2 will be assessed at baseline (enrollment).
  Activation of the inactive prothrombin to the active thrombin will be estimated from concentrations of prothrombin fragment 1 + 2 (pmol/L), using a commercial enzyme-linked immunosorbent assay (ELISA). Prothrombin fragment 1 + 2 are the byproducts of the abovementioned activation process.

SECONDARY OUTCOMES:
Levels of von Willebrand factor (vWF) antigen | von Willebrand factor antigen will be assessed at baseline (enrollment).
  von Willebrand factor plays an important role in platelet plug formation and will be one of the secondary outcome measures. von Willebrand factor antigen (%) will be measured using an in-house immunoassay.
Concentration of cleaved high-molecular weight kininogen (cHK) | cHK will be assessed at baseline (enrollment).
  cHK is an essential component of the contact activation system of the coagulation cascade. cHK (µg/ml) will be measured with the help of enzyme-linked immunosorbent assay (ELISA).
Concentration of coagulation factor XII (FXII) | FXII will be assessed at baseline (enrollment).
  FXII is an essential component of the contact activation system of the coagulation cascade. FXII (µg/ml) will be measured with the help of enzyme-linked immunosorbent assay (ELISA).
Concentration of prekallikrein | Prekallikrein will be assessed at baseline (enrollment).
  Prekallikrein is an essential component of the contact activation system of the coagulation cascade. Prekallikrein (µg/ml) will be measured with the help of enzyme-linked immunosorbent assay (ELISA).
Concentration of high-molecular weight kininogen (HK) | HK will be assessed at basline (enrollment).
  HK plays a key role in the contact activation system of the coagulation cascade. HK (%) will be measured using enzyme-linked immunosorbent assay (ELISA).
Concentration of C1-inhibitor | C1-inhibitor will be assessed at baseline (enrollment).
  C1-inhibitor is the main regulator of the contact activation system. Concentration of C1-inhibitor (g/L) will be measured using nephelometry.
Concentration of coagulation factor VII (FVII) | FVII will be assessed at baseline (enrollment).
  FVII plays an important role in the secondary hemostasis. Concentration of FVII (%) will be measured using clot assay.
Concentration of coagulation factor X (FX) | FX will be assessed at baseline (enrollment).
  FX plays an important role in the secondary hemostasis. Concentration of FX (%) will be measured using clot assay.
Concentration of coagulation factor II (FII) | FII will be assessed at baseline (enrollment).
  FII plays an important role in the secondary hemostasis. Concentration of FII (%) will be measured using clot assay.
Concentration of protein C | Protein C will be assessed at baseline (enrollment).
  Protein C is essential for the regulation of the blood coagulation cascade. Concentration of protein C (%) will be measured using chromogenic assay.
Concentration of protein S | Protein S will be assessed at baseline (enrollment).
  Protein S is essential for the regulation of the blood coagulation cascade. Concentration of protein S (%) will be measured using turbidity.
Concentration of antithrombin (AT). | Antithrombin will be assessed at baseline (enrollment).
  Antithrombin is essential for the regulation of the blood coagulation cascade. Concentration of antithrombin (%) will be measured using chromogenic assay.
Concentration of tissue factor pathway inhibitor (TFPI) | TFPI will be assessed at baseline (enrollment).
  TFPI is important in the regulation of the blood coagulation system. TFPI (pg/ml) will be measured using enzyme-linked immunosorbent assay (ELISA).
Fibrin turnover assessed by maximum lysis velocity (Vmax) | Fibrin turnover, assessed by Vmax, will be measured at baseline (enrollment).
  Fibrin turnover will be assessed through fibrin clot lysis, where measurement of Vmax (optical density (OD)/min) will be conducted.
Fibrin turnover assessed by peak optical density (OD) | Fibrin turnover, assessed by peak OD, will be measured at baseline (enrollment).
  Fibrin turnover will be assessed through fibrin clot lysis, where measurement of peak OD (OD) will be conducted.
Fibrin turnover assessed by clot lysis | Fibrin turnover, assessed by clot lysis, will be measured at baseline (enrollment).
  Fibrin turnover will be assessed through fibrin clot lysis, where measurement of clot lysis (%) will be conducted.
Fibrin turnover assessed by overall hemostatic potential (OHP) | Fibrin turnover, assessed by OHP, will be measured at baseline (enrollment).
  Fibrin turnover will be assessed through fibrin clot lysis, where measurement of OHP (OD x min) will be conducted.
Fibrin turnover assessed by fiber diameter | Fibrin turnover, assessed by fiber diameter, will be measured at baseline (enrollment).
  Fibrin turnover will be assessed through fibrin clot lysis, where measurement of fiber diameter (µm) will be conducted.
Fibrin turnover assessed by fiber density | Fibrin turnover, assessed by fiber density, will be measured at baseline (enrollment).
  Fibrin turnover will be assessed through fibrin clot lysis, where measurement of fiber density (x 10^6 Da/cm^3) will be conducted.
Concentration of fibrinogen | Fibrinogen will be assessed at baseline (enrollment).
  Conversion of fibrinogen to fibrin, in which thrombin plays a key role, is essential for blood coagulation. Concentrations of fibrinogen (µmol/L) will be measured using nephelometry.
Concentration of D-dimer | D-dimer will be assessed at baseline (enrollment).
  D-dimer is a fibrin degradation product that reflects the fibrinolysis process (the breakdown of fibrin network), which plays a crucial role in preventing blood clots from causing complications. D-dimer (mg/L) will be measured using immunoassay.
Concentration of tissue-type plasminogen activator (t-PA) | t-PA will be assessed at baseline (enrollment).
  t-PA is a protein that stimulates the breakdown of blood clots. It helps convert plasminogen into its active form, plasmin, the major enzyme responsible for the breakdown of blood clots. Concentration of t-PA (ng/ml) will be measured using enzyme-linked immunosorbent assay (ELISA).
Concentration of plasminogen activator inhibitor 1 (PAI-1) | PAI-1 will be assessed at baseline (enrollment).
  PAI-1 functions as the inhibitor of t-PA, which will stimulate the formation of blood clots. Concentration of PAI-1 (ng/ml) will be measured using enzyme-linked immunosorbent assay (ELISA).
Levels of plasminogen | Plasminogen will be assessed at baseline (enrollment).
  Plasminogen is the inactive form of plasmin, the major enzyme that breaks down blood clots. Levels of plasminogen (%) will be measured using chromogenic assay.
Levels of coagulation factor XIII (FXIII) | FXIII will be assessed at baseline (enrollment).
  FXIII plays a key role in stabilizing the blood clots. Levels of FXIII will be measured using immunoassay.
Levels of plasmin inhibitor (PI) | PI will be assessed at baseline (enrollment).
  PI is the major inhibitor of plasmin. Levels of PI (%) will be measured using chromogenic assay.
Levels of thrombin activatable fibrinolysis inhibitor (TAFI) | TAFI will be assessed at baseline (enrollment).
  TAFI is an enzyme that is activated by thrombin, which downregulates fibrinolysis, stimulating blood clot formation. Levels TAFI will be measured using enzyme-linked immunosorbent assay (ELISA).
Assessment of atrial fibrillation burden (AF-burden) | AF-burden will be assessed from baseline (enrollment) to the end of heart rhythm monitoring at seven days.
  AF-burden is associated with stroke, making it an important factor in the treatment of atrial fibrillation. AF-burden (%) will be determined as a percentage, based on the total number of atrial fibrillation events during the seven days heart rhythm monitoring.
Assessment of left atrial function index (LAFI) | LAFI will be assessed at baseline (enrollment).
  Using cardiac ultrasound, also known as echocardiography, a rhythm independent expression of left atrial function, known as LAFI, will be assessed. Left atrial function has been proven to modify the risk of stroke in patients with atrial fibrillation. LAFI (cm/ml/m^2) will be given as a numerical value, with higher numbers indicating better left atrial function.
Assessment of underlying heart failure with preserved ejection fraction (HFpEF) using the HFA-PEFF score | HFpEF will be assessed at baseline (enrollment).
  HFpEF is characterized by abnormal diastolic function, which corresponds to an increase in the stiffness of the heart. The HFA-PEFF score will be used in the assessment of underlying HFpEF. The HFA-PEFF score ranges from 0-6 points, with a score of ≥ 5 considered to be diagnostic of HFpEF.
Assessment of underlying heart failure with preserved ejection fraction (HFpEF) using the H2FPEF score | HFpEF will be assessed at baseline (enrollment).
  HFpEF is characterized by abnormal diastolic function, which corresponds to an increase in the stiffness of the heart. The H2FPEF score will be used in the assessment of underlying HFpEF. The H2FPEF score ranges from 0-9 points, with a score of ≥ 6, associated with a high probability of HFpEF.

CONTACTS AND LOCATIONS:
Locations (1):
- Esbjerg Hospital - University Hospital of Southern Denmark, involving collaboration between the Unit for Thrombosis Research, Department of Clinical Diagnostics and the Department of Cardiology., Esbjerg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
It is too preliminary, at this stage; however, investigators do not rule out the possibility of sharing individual participant data (IPD) in the future.

REFERENCES:
- [Background] Ariyaratnam JP, Mishima RS, Kadhim K, Emami M, Fitzgerald JL, Thiyagarajah A, Dziano JK, Howie JO, Middeldorp ME, Sanders P, Elliott AD. Utility and Validity of the HFA-PEFF and H2FPEF Scores in Patients With Symptomatic Atrial Fibrillation. JACC Heart Fail. 2024 Jun;12(6):1015-1025. doi: 10.1016/j.jchf.2024.01.015. Epub 2024 Mar 20. PMID 38520461
- [Background] Thomas L, Hoy M, Byth K, Schiller NB. The left atrial function index: a rhythm independent marker of atrial function. Eur J Echocardiogr. 2008 May;9(3):356-62. doi: 10.1016/j.euje.2007.06.002. Epub 2007 Aug 7. PMID 17689293
- [Background] Glowicki B, Matusik PT, Plens K, Undas A. Prothrombotic State in Atrial Fibrillation Patients With One Additional Risk Factor of the CHA2DS2-VASc Score (Beyond Sex). Can J Cardiol. 2019 May;35(5):634-643. doi: 10.1016/j.cjca.2019.01.014. Epub 2019 Jan 30. PMID 30955928
- [Background] Ding WY, Gupta D, Lip GYH. Atrial fibrillation and the prothrombotic state: revisiting Virchow's triad in 2020. Heart. 2020 Oct;106(19):1463-1468. doi: 10.1136/heartjnl-2020-316977. Epub 2020 Jul 16. PMID 32675218
- [Background] Tilly MJ, Geurts S, Pezzullo AM, Bramer WM, de Groot NMS, Kavousi M, de Maat MPM. The association of coagulation and atrial fibrillation: a systematic review and meta-analysis. Europace. 2023 Feb 8;25(1):28-39. doi: 10.1093/europace/euac130. PMID 35942591
- [Background] Benz AP, Hijazi Z, Lindback J, Connolly SJ, Eikelboom JW, Oldgren J, Siegbahn A, Wallentin L. Biomarker-Based Risk Prediction With the ABC-AF Scores in Patients With Atrial Fibrillation Not Receiving Oral Anticoagulation. Circulation. 2021 May 11;143(19):1863-1873. doi: 10.1161/CIRCULATIONAHA.120.053100. Epub 2021 Apr 14. PMID 33849281
- [Background] Hijazi Z, Lindback J, Alexander JH, Hanna M, Held C, Hylek EM, Lopes RD, Oldgren J, Siegbahn A, Stewart RA, White HD, Granger CB, Wallentin L; ARISTOTLE and STABILITY Investigators. The ABC (age, biomarkers, clinical history) stroke risk score: a biomarker-based risk score for predicting stroke in atrial fibrillation. Eur Heart J. 2016 May 21;37(20):1582-90. doi: 10.1093/eurheartj/ehw054. Epub 2016 Feb 25. PMID 26920728
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550